CLINICAL TRIAL: NCT02676349
Title: Two Arm, Prospective, Multicenter Randomized Phase II Trial of Neoadjuvant Modified Folfirinox Regimen, With or Without Preoperative Concomitant Chemoradiotherapy in Patients With Borderline Resectable Pancreatic Carcinoma
Brief Title: Neoadjuvant mFolfirinox With or Without Preoperative Concomitant Chemoradiotherapy in Patients With Borderline Resectable Pancreatic Carcinoma (PANDAS-PRODIGE 44)
Status: Active, not recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Institut de Cancérologie de Lorraine (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2014-005681-29
Record Dates: First submitted 2016-02-03; First posted 2016-02-08 (Estimated); Last update posted 2023-09-28 (Actual); Status verified 2023-09

CONDITIONS: Pancreatic Carcinoma
Keywords: mFolfirinox; Chemoradiotherapy; Neoadjuvant treatment; Borderline
MeSH Terms: conditions — Pancreatic Neoplasms | interventions — Chemoradiotherapy; Surgical Procedures, Operative; Chemotherapy, Adjuvant

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Arm B (Experimental): Neoadjuvant chemotherapy with mFolfirinox regimen + concomitant chemoradiotherapy + surgery + adjuvant chemotherapy
  Interventions: Drug: mFolfirinox; Radiation: Chemoradiotherapy; Procedure: surgery; Drug: Adjuvant chemotherapy
- Arm A (Active Comparator): Neoadjuvant chemotherapy with mFolfirinox regimen + surgery + adjuvant chemotherapy
  Interventions: Drug: mFolfirinox; Procedure: surgery; Drug: Adjuvant chemotherapy

INTERVENTIONS:
Drug: mFolfirinox — oxaliplatin folinic acid irinotecan 5FU oxaliplatin
Radiation: Chemoradiotherapy — conformational external irradiation (50.4 Gy) + capecitabine
  Arms: Arm B
Procedure: surgery — 1 to 4 weeks after neoadjuvant treatment according to tumour response
Drug: Adjuvant chemotherapy — Gemcitabine or modified LV5FU (folinic acid+-bolus fluorouracil+ infusional fluorouracil)

SUMMARY:
This is a prospective, randomized phase II trial. The aim of this study is to assess the efficacy of two therapeutics strategies. Patients with borderline-resectable pancreatic cancer (BRPC) will be randomly in two arms : neoadjuvant mFolfirinox followed with or without preoperative chemoradiotherapy with capecitabine.

DETAILED DESCRIPTION:
Surgery, especially if followed by adjuvant chemotherapy, offers the only chance of cure of pancreatic cancer. At first diagnosis, after careful assessment, only 10 to 15% of patients are considered to be candidates for surgical resection and about 7% have a potentially resectable disease. These potentially resectable tumors called "borderline resectable pancreatic cancer" (BRPC) are conceptualized as those that involve the mesenteric vasculature to a limited extent and those for which resection, while possible, would likely be compromised by positive surgical margins (R1) in the absence of neoadjuvant treatment. R0 resection is indeed considered as an independent prognostic factor for survival when the surgical procedures, histological examination and definition of microscopic invasion are standardized.

The objectives of neoadjuvant treatments of BRPC is to reduce tumor volume before surgery in order to improve the chances of radical (R0) resection and to reduce the rate of lymph node positivity and recurrences. The primary outcome in published studies is usually R0 resection rate, but these results also depend on the number of margins examined and the definition of microscopic margin involvement. Prospective studies with consistent selection criteria and standardized assessment criteria are needed.

Different neoadjuvant therapeutic strategies have been tested in pilot studies: preoperative chemoradiotherapy or neoadjuvant chemotherapy, followed or not by a preoperative (chemo)radiotherapy. Due to the lack of randomized studies, the best sequence of treatment administration has not been established.

The aim of this prospective, randomized, multicenter, trial is to evaluate the R0 resection rate with neoadjuvant Folfirinox, followed or not by radiochemotherapy for patients with borderline resectable pancreatic cancers.

ELIGIBILITY:
Inclusion Criteria:

* ECOG performance status 0 or 1
* Adult patients ≥ 18 years and ≤ 75 years of age
* Histologic or cytologic proven adenocarcinoma of the pancreas (histologic confirmation of diagnosis is preferred)
* Confirmation by independent multidisciplinary expert review of borderline resectable status, according to NCCN-Clinical Practice Guidelines in Oncology "pancreatic adenocarcinoma", version 1.2015.
* Adequate hematologic function, as follows:
* absolute neutrophil count (ANC) ≥ > 2000/mm3
* platelet count ≥ 100 000/mm3
* haemoglobin ≥ 10 g/dL
* Adequate renal, hepatic and bone marrow function, defined as:

  * Calculated creatinine clearance ≥ 50 mL/min according to MDRD formula
  * Serum total bilirubin ≤ 1.5 times the institutional upper limit of normal. Patients with a biliary short metal stent due to cancer obstruction may be included provided that high-quality imaging is performed before stenting and bilirubin level after stent insertion decreased to ≤ 20 mg/L (≤ 34 µmol/l), and there is no cholangitis.
* Male and female subjects who agree to use highly effective methods of birth control (e.g., condoms, combined oral contraceptives, some intrauterine devices [IUDs], sexual abstinence, or sterilized partner)

  * for male subject: during the treatment and for up to 6 months after the last dose of oxaliplatin or up to 3 months after the last dose of irinotcan.
  * for female subject: during the treatment and for up to 4 months after the last dose of oxaliplatin or up to 3 months after the last dose of irinotcan.
* Ability to provide written informed consent before the start of any study specific procedures
* Patient's legal capacity to consent to study participation and to understand and comply with the requirements of the study.

Exclusion Criteria:

* Any previous treatment of the pancreatic cancer except biliary short metal stenting (chemotherapy, targeted tumor therapy, local ablative therapy, previous irradiation within the actual fields of planned radiotherapy)
* Evidence of distant metastases including ascites
* Evidence of extent of pancreatic cancer beyond that defined as "borderline resectable" : suspicious lymphadenopathy outside of the standard field of resection (i.e., aortocaval nodes, distant abdominal nodes)
* Contraindication for pancreas resection
* Pregnant or breast feeding females
* Patients with known Gilbert's Syndrome or homozygosity for UGT1A1*28 polymorphism
* Uracilemia ≥ 16ng/mL either a partial or complete deficiency in dihydropyrimidine dehydrogenase (DPD)
* Participation in any other clinical trial or treatment with any experimental drug within 28 days before enrolment to the study or during study participation until the end of treatment visit that can be interfering with the objectives of the study
* Previous or concurrent malignant tumor disease other than underlying tumor disease (with the exception of cervical cancer in situ, adequately treated non-melanoma skin cancers, superficial bladder tumors (Ta, Tis, and T1) or any curatively treated without chemotherapy and favourable prognosis tumors without evidence of disease for > 3 years prior to enrolment)
* Any severe and/or uncontrolled medical conditions including but not limited to:

  * Clinically significant cardiovascular or vascular disease : angina pectoris (even controlled), previous myocardial infarction, serious uncontrolled cardiac arrhythmia, chronic heart failure, acute or chronic infectious disease requiring general treatment)
  * Acute and chronic, active infectious disorders that requires systemic treatment
  * Peripheral polyneuropathy > grade 1
  * Any previous inflammatory disease of colon or rectum
  * Any other severe concomitant disease or disorder, which could influence patient's ability to participate in the study and his/her safety during the study e.g. severe hepatic, renal, pulmonary, metabolic, or psychiatric disorders
* Uncorrected disturbed electrolyte balance, in particular hypokalemia or hypocalcemia
* Hypersensitivity against any of the study drugs (gemcitabine, oxaliplatin, irinotecan, 5-fluorouracil, folinic acid), or the ingredients of these drugs (e.g. fructose).

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 130 (Actual)
Dates: Start 2016-10-13 (Actual); Primary Completion 2024-06 (Estimated); Study Completion 2027-10 (Estimated)

PRIMARY OUTCOMES:
To assess the efficacy of two neoadjuvant therapies in patients with borderline resectable pancreatic carcinoma evaluated on histological R0 resection margin rate | up to 7.5 months

SECONDARY OUTCOMES:
Evaluate the toxicities associated with chemotherapy and chemoradiotherapy | up to 7 years
Evaluate the proportion of resected patients | up to 7.5 months
Evaluate the response rate to chemotherapy and chemoradiotherapy | up to 7.5 months
Evaluate the histological complete response rate in resected patients. | up to 7.5 months
Evaluate the perioperative mortality rate | up to 8.5 months
Evaluate the perioperative morbidity rate | up to 8.5 months
Evaluate the overall survival | up to 7 years
Evaluate the quality of life | up to 7.5 months
Evaluate the loco-regional relapse-free survival | 7 years
Evaluate the metastatic Progression Free Survival | 7 years
Evaluate the progression-free survival | 7 years

CONTACTS AND LOCATIONS:
Overall Officials: Thierry CONROY, Pr, Principal Investigator — Institut de Cancérologie de Lorraine; Jean-Baptiste BACHET, Pr, Study Chair — Groupe Hospitalier Pitié-Salpêtrière; Pascal HAMMEL, Pr, Study Chair — Hôpital Paul Brousse - Hôpitaux de Paris (AP-HP)
Locations (26):
- France (26):
  - Institut Bergonié, Bordeaux
  - Polyclinique Bordeaux Nord, Bordeaux
  - Hôpital Beaujon, Clichy
  - Chu Colmar, Colmar
  - Hôpital Henri Mondor (APHP), Créteil
  - Centre Oscar Lambret, Lille
  - Chru Lille, Lille
  - Infirmerie Protestante de Lyon, Lyon
  - Hôpital Européen Marseille, Marseille
  - Hôpital La Timone, Marseille
  - Institut Paoli CALMETTES, Marseille
  - Institut du Cancer de Montpellier, Montpellier
  - Chu Nantes, Nantes
  - Hôpital Cochin (APHP), Paris
  - Institut Mutualiste Montsouris, Paris
  - Pitié Salpêtrière (APHP), Paris
  - Hôpital Haut-Lévêque, Pessac
  - CHU Reims, Reims
  - Centre Eugène Marquis, Rennes
  - Chu Rouen, Rouen
  - CHP Saint Grégoire, Saint-Grégoire
  - Institut de Cancérologie de l'Ouest, Saint-Herblain
  - Chru Tours, Tours
  - Chru Nancy, Vandœuvre-lès-Nancy
  - Institut de Cancérologie de Lorraine, Vandœuvre-lès-Nancy
  - Hôpital Paul Brousse, Villejuif

IPD SHARING:
Plan to Share IPD: No